CLINICAL TRIAL: NCT00923247
Title: A Targeted Ph I/II Trial of ZD6474 (Vandetanib; CAPRELSA) Plus the Proteasome Inhibitor, Bortezomib (Velcade ), in Adults With Solid Tumors With a Focus on Hereditary or Sporadic, Locally Advanced or Metastatic Medullary Thyroid Ca (MTC)
Brief Title: A Targeted Phase I/II Trial of ZD6474 (Vandetanib; ZACTIMA) Plus the Proteasome Inhibitor, Bortezomib (Velcade ), in Adults With Solid Tumors With a Focus on Hereditary or Sporadic, Locally Advanced or Metastatic Medullary Thyroid Cancer (MTC)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Terminated due to slow accrual,primary endpoint reached & investigator left NIH.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ravi A. Madan, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 090089; 09-C-0089; NCT00863720 (obsolete NCT alias)
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Results first posted 2017-05-17 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Medullary Thyroid Carcinoma
Keywords: Vandetanib; Bortezomib; Medullary Thyroid; Proteasome Inhibitor; Cancer; Solid Tumor; Thyroid Cancer; Medullary Thyroid Cancer
MeSH Terms: conditions — Carcinoma, Medullary; Neoplasms; Thyroid Neoplasms | interventions — Bortezomib; vandetanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1 - vandetanib and bortezomib (Experimental): Patients will be treated with vandetanib and bortezomib to find the maximally tolerated dose
  Interventions: Drug: Bortezomib; Drug: Vandetanib
- Phase 2 B - vandetanib alone (Active Comparator): Patients will be treated with vandetanib alone.
  Interventions: Drug: Vandetanib
- Phase 2 A - vandetanib and bortezomib at the MTD (Active Comparator): Patients will be treated with vandetanib and bortezomib at the maximally tolerated dose (MTD) of the Phase I study
  Interventions: Drug: Bortezomib; Drug: Vandetanib

INTERVENTIONS:
Drug: Bortezomib — This study is designed to assess the safety, tolerance and activity of daily oral vandetanib and bortezomib on days 1, 4, 8 & 11 every 28 days in adults
  Other Names: Velcade
  Arms: Phase 1 - vandetanib and bortezomib; Phase 2 A - vandetanib and bortezomib at the MTD
Drug: Vandetanib — This study is designed to assess the safety, tolerance and activity of daily oral vandetanib and bortezomib on days 1, 4, 8 & 11 every 28 days in adults
  Other Names: Caprelsa

SUMMARY:
Background:

* The combination of anti-cancer drugs vandetanib (given orally) and bortezomib (given intravenously) has not been used in humans. However, both drugs have been studied separately. Bortezomib has been approved by the U.S. Food and Drug Administration (FDA) for treating multiple myeloma and mantle cell lymphoma, while vandetanib is still under investigation pending FDA approval.
* Both bortezomib and vandetanib are under investigation for use in treating certain kinds of cancer. Researchers hope that the combination of these two drugs will be more effective than either of them alone.

Objectives:

* To determine if the combination of vandetanib and bortezomib will decrease the amount of the cancer and, if it does, to determine how long the response will last.
* To determine any side effects that may occur with this combination of treatments.
* To determine what doses of each drug are well tolerated and safe when given together.
* To study genetic mutations in tumors to better understand how tumors grow and how these drugs interact with the tumor.

Eligibility:

* Patients 18 years of age and older with solid tumors that cannot be surgically removed and have either recurred or shown further growth. The tumor(s) must be able to be evaluated by X-ray, MRI (magnetic resonance imaging), and CT (computerized tomography) scanning.
* Patients who have been diagnosed with medullary thyroid cancer will participate in Phase II of the study.

Design:

* Tumor samples may be taken at the start of the study for research purposes.
* Phase I: Patient groups will be treated on an outpatient basis with vandetanib and bortezomib, given at increasing doses over four different levels to determine the maximum tolerated dose calculated by height and weight:
* Doses will be given on Days 1, 4, 8, and 11 for each 28-day cycle.
* Two additional levels (Level 1A and Level 1B) may be included in the study, depending on side effects at various levels.
* Phase II: Patients with medullary thyroid cancer will be divided into two groups, with two patients in Group A for every one patient in Group B. No placebo will be involved in this study.
* Group A: Patients will be treated with vandetanib and bortezomib at the maximally tolerated dose of the Phase I study.
* Group B: Patients will be treated with bortezomib alone.
* A second tumor sample may be taken. In patients with thyroid cancer, the second biopsy will be done at the 6-week evaluation (approximately 42 days after beginning). In patients with cancer other than thyroid cancer, the second biopsy will be obtained on Day 4 of either the first or second cycle, after the bortezomib infusion.
* The effects of the drugs will be studied through blood samples and CT scans taken during and after various drug cycles.

DETAILED DESCRIPTION:
Background:

* Vandetanib (CAPRELSA; ZD6474) potently inhibits vascular endothelial growth factor receptor-2 (VEGFR-2), and shows additional inhibitory activity at sub-micromolar concentrations against the Rearranged during Transfection (RET) receptor, Flt-4 and EGF receptor tyrosine kinases.
* Clinical trials have shown that vandetanib is active against medullary thyroid carcinomas (MTCs), but the activity is characterized by partial responses of variable duration, underscoring the need to develop active combinatorial regimens.
* Bortezomib (PS-341, Velcade ), a proteasome inhibitor, has been reported to have several putative mechanisms of action and it is likely that its toxicity is mediated by affecting more than one pathway or target. Bortezomib is reported to inhibit the nuclear factor kappa-light-chain-enhancer of activated B cells (NF-kappaB) pathway and regulate NF-kappaB-dependent expression of several other inhibitors of apoptosis.
* In vitro studies have shown bortezomib to be active against a broad range of thyroid cancer cell lines. Given this activity of bortezomib and the role of the proteasome in regulating diverse cellular pathways, this study proposes to combine bortezomib with vandetanib to treat patients with advanced solid tumors with a focus on patients with MTC.

Objectives:

* To assess the activity of vandetanib plus bortezomib in adults with MTC, using Response Evaluation Criteria in Solid Tumors (RECIST) and tumor biomarkers including carcinoembryonic antigen (CEA) and calcitonin as endpoints.
* To assess the safety and tolerance of vandetanib plus bortezomib in dose-seeking cohorts.
* To compare the combination bortezomib plus vandetanib versus vandetanib alone in adults with MTC by assessing the response rate and progression-free survival
* In exploratory analyses: (a) examine the correlation between genotype and response to therapy in patients with MTC, (b) examine the extent, if any, of rearranged during transfection (RET) inhibition in patients with MTC following the administration of vandetanib; and (c) examine the effect, if any, of bortezomib on microtubules.

Eligibility:

* Adults age 18 and older with unresectable, recurrent or metastatic solid tumors, including MTC.
* Disease must be evaluable by RECIST.

Design:

* Phase I dose-escalation study followed by randomized phase II trial.
* Maximum total number for planned enrollment: 117 - Dose-seeking cohorts of three to 6 patients until maximum tolerated dose (MTD)/dose limiting toxicity (DLT) reached (up to 24 patients) followed by a randomized phase II trial comparing the activity of the combination of bortezomib plus vandetanib with vandetanib alone (2:1 randomization 62 plus 31 equals 93 patients).
* The MTD and DLT will be determined based on toxicities during the first eight weeks of combined therapy.
* Cycle length will be four weeks. Response will be determined by RECIST every 12 weeks.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Pathologic confirmation of cancer by the Laboratory of Pathology, National Cancer Institute (NCI)
2. Phase I: Diagnosis of recurrent, metastatic or primary unresectable solid tumor that does not have curative standard treatment.

   Phase II: Diagnosis of recurrent, metastatic or primary unresectable medullary thyroid cancer (MTC).
3. Measurable disease at presentation: Either by Response Evaluation Criteria in Solid Tumors (RECIST) or by measurement of serum markers (calcitonin, carcinoembryonic antigen (CEA), prostate specific antigen (PSA) or cancer antigen 125 or carbohydrate antigen 125 (CA-125) in the dose-finding portion of the study; with disease measurable by RECIST required only in the phase II cohort.
4. A life expectancy of at least 3 months and Eastern Cooperative Oncology Group (ECOG) performance status 0 1.
5. Age greater than or equal to 18 years
6. Last dose of chemotherapy or experimental therapy more than 4 weeks (6 weeks in the case of nitrosourea) prior to enrollment date; unless the last therapy consisted of an oral agent whose average half life is known to be less than 48 hours in which case only 2 weeks need to have elapsed. Regardless of the therapy, any toxicity greater than Common Terminology Criteria in Adverse Events (CTCAE) grade 1 from previous anti-cancer therapy must have been resolved.
7. Last radiotherapy treatment 4 weeks prior to starting treatment with this protocol with the exception of palliative radiotherapy and there must be sites of measurable disease that did not receive radiation.
8. Organ and marrow function as defined:

   * total bilirubin less than 1.5 times the upper limit of reference range (ULRR), unless the patient meets the criteria for Gilbert's Syndrome
   * alanine aminotransferase (ALT), aspartate aminotransferase (AST) and alkaline phosphatase (ALP) all three less than 2.5 times the upper limit of the reference range (ULRR), or less than 5 times the ULRR if judged by the investigator to be related to liver metastases
   * serum creatinine less than 1.5 times the ULRR or creatinine clearance greater than or equal to 30 mL/minute (calculated by Cockcroft-Gault formula or measured in a timed urine collection)
   * serum calcium below the CTCAE grade 1 upper limit (11.5mg/dL or 2.9 mmol/L). In cases where the serum calcium is below the normal range, the calcium adjusted for albumin is calculated and substituted for the measured value.
   * serum potassium greater than the lower limit of normal (LLN) and less than 5.5 mmol/L.
   * serum magnesium greater than the LLN and less than 3.0 mg/dL or 1.23 mmol/L.
   * absolute neutrophil count greater than or equal to 1000/mm(3)
   * platelet count greater than or equal to 100,000/mm(3)
   * Prothrombin time (PT) less than or equal to 4 seconds above ULN and partial thromboplastin time (PTT) less than or equal to 10 seconds above ULN.
9. Ability to understand and sign an informed consent document.
10. Provision of informed consent prior to any study-related procedures
11. Negative pregnancy test for women of childbearing potential
12. Ability and willingness to follow the guidelines of the clinical protocol including visits to National Cancer Institute (NCI), Bethesda, Maryland for treatment and follow up visits.
13. Because the effects of chemotherapy on the developing human fetus are potentially harmful, female patients must be one year post-menopausal, surgically sterile, or using an acceptable method of contraception during and continued after the last dose of study medications (oral contraceptives, barrier methods, approved contraceptive implant, long-term injectable contraception, intrauterine device or tubal ligation). Male patients must be surgically sterile or using an acceptable method of contraception during their participation in this study. Contraceptive use will continue for at least four months after the last dose of study medication.

EXCLUSION CRITERIA:

1. Patients with cancer potentially curable by surgical excision alone or patients who have not received therapy that might be considered standard and potentially curable.
2. Evidence of severe or uncontrolled systemic disease or any concurrent condition including, but not limited to symptomatic congestive heart failure, unstable angina pectoris, unstable hypertension, seizure disorder, or psychiatric illness which in the Investigators opinion makes it undesirable for the patient to participate in the trial or which would jeopardize compliance with the protocol.
3. Untreated brain metastases (or local treatment of brain metastases within the last 6 months) due to the poor prognosis of these patients and difficulty ascertaining the cause of neurologic toxicities.
4. During Phase II enrollment: Prior therapy with vandetanib.
5. Women who are currently pregnant or breast-feeding, due to the possible adverse effects on the developing fetus and infants.
6. The presence of a second malignancy within the last 2 years, other than squamous cell carcinoma of the skin or in situ cervical cancer because it will complicate the primary objective of the study. Cancer survivors who have been free of disease for at least two years can be enrolled in this study.

   - There is one other exception to the exclusion of secondary malignancies: multiple endocrine neoplasia type 2 (MEN2) patients with concurrent medullary thyroid cancer and pheochromocytoma may be enrolled at the discretion of the Principal Investigator.
7. Patients with evidence of a bleeding diathesis that cannot be corrected with standard therapy or factor replacement.
8. Any unresolved toxicity greater than CTCAE grade 1 (except alopecia) from previous anticancer therapy. Patients with grade 1 neuropathy will be evaluated on a case by case basis for entry into study. Baseline conditions will be taken into consideration.
9. Major surgery within 4 weeks, or incompletely healed surgical incision before starting study therapy.
10. Clinically significant cardiovascular event (e.g. myocardial infarction, superior vena cava syndrome (SVC), New York Heart Association (NYHA) classification of heart disease greater than or equal to 2 within 3 months before entry; or presence of cardiac disease that, in the opinion of the Investigator, increases the risk of ventricular arrhythmia.
11. History of arrhythmia (multifocal premature ventricular contractions PVCs, bigeminy, trigeminy, ventricular tachycardia, or uncontrolled atrial fibrillation) which is symptomatic or requires treatment (CTCAE grade 3) or asymptomatic sustained ventricular tachycardia. Atrial fibrillation controlled on medication is not excluded.
12. History (within the last 6 months) or presence of stroke/cerebrovascular accident.
13. Corrected QT interval (QTc) prolongation with other medications. If the medication can be discontinued and an alternative medication started that does not cause QTc prolongation, the patient would be eligible. If no alternative medication is available and the medication cannot be discontinued for medical reasons, then the patient would not be eligible.
14. Congenital long Q wave, T wave (QT) syndrome, or 1st degree relative with unexplained sudden death under 40 years of age.
15. Presence of left bundle branch block (LBBB).
16. QTc with Bazett's correction that is not measurable, or greater than or equal to 480 msec on screening electrocardiogram (ECG). (Note: If a patient has a QTc interval greater than or equal to 480 msec on screening ECG, the screen ECG may be repeated twice (at least 24 hours apart). The average QTc from the three screening ECGs must be less than 480 msec in order for the patient to be eligible for the study). Patients who are receiving a drug that has a risk of QTc prolongation are excluded if QTc is greater than or equal to 460 msec.
17. Concurrent medication that may cause QTc prolongation or induce Torsades de Pointes: Those medications in Group One will not be allowed. Those medications in Group Two will be allowed.
18. Hypertension not controlled by medical therapy (systolic blood pressure greater than 160 mm Hg or diastolic blood pressure greater than 100 mm Hg)
19. Currently active (uncontrolled) diarrhea greater than or equal to CTCAE Grade 2 that may affect the ability of the patient to absorb the vandetanib or tolerate diarrhea. Antidiarrhea medications are allowed in patients with chronic diarrhea.
20. Concomitant medications that are potent inducers (rifampicin, rifabutin, phenytoin, carbamazepine, phenobarbital and St. John's Wort) of cytochrome P450 3A4 (CYP3A4) function.
21. Major surgery within 4-weeks, or incompletely healed surgical incision before starting study medications. Biopsies, port placements, and dental work are examples of acceptable (nonmajor) surgery within the 4 week time frame.
22. Inability to take oral medications for whatever reason.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-02-19 (Actual); Primary Completion 2016-04-01 (Actual); Study Completion 2016-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ravi A Madan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davies L, Welch HG. Increasing incidence of thyroid cancer in the United States, 1973-2002. JAMA. 2006 May 10;295(18):2164-7. doi: 10.1001/jama.295.18.2164. PMID 16684987
- [Background] Truong T, Rougier Y, Dubourdieu D, Guihenneuc-Jouyaux C, Orsi L, Hemon D, Guenel P. Time trends and geographic variations for thyroid cancer in New Caledonia, a very high incidence area (1985-1999). Eur J Cancer Prev. 2007 Feb;16(1):62-70. doi: 10.1097/01.cej.0000236244.32995.e1. PMID 17220706
- [Background] Burgess JR, Tucker P. Incidence trends for papillary thyroid carcinoma and their correlation with thyroid surgery and thyroid fine-needle aspirate cytology. Thyroid. 2006 Jan;16(1):47-53. doi: 10.1089/thy.2006.16.47. PMID 16487013
- [Result] Abstract: Phase I/II trial of vandetanib and bortezomib in adults with locally advanced or metastatic medullary thyroid cancer: Phase I results. A. W. Gramza, S. A. Wells, S. Balasubramaniam, and A. T. Fojo Journal of Clinical Oncology 2011 29:15_suppl, 5565-5565
- [Derived] Del Rivero J, Edgerly M, Ward J, Madan RA, Balasubramaniam S, Fojo T, Gramza AW. Phase I/II Trial of Vandetanib and Bortezomib in Adults with Locally Advanced or Metastatic Medullary Thyroid Cancer. Oncologist. 2019 Jan;24(1):16-e14. doi: 10.1634/theoncologist.2018-0452. Epub 2018 Oct 8. PMID 30297385
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2009-C-0089.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No participants were enrolled in the phase IIB cohort.
Groups:
- Phase 1 - Vandetanib and Bortezomib: Patients will be treated with vandetanib and bortezomib to find the maximally tolerated dos
  Bortezomib: This study is designed to assess the safety, tolerance and activity of daily oral vandetanib and bortezomib on days 1, 4, 8 & 11 every 28 days in adults
  Vandetanib: This study is designed to assess the safety, tolerance and activity of daily oral vandetanib and bortezomib on days 1, 4, 8 & 11 every 28 days in adults
Period: Overall Study
Arm/Group | Phase 1 - Vandetanib and Bortezomib | Phase 2 A - Vandetanib and Bortezomib at the MTD
Started | 21 | 1
Completed | 21 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase 1: Patients will be treated with vandetanib and bortezomib to find the maximally tolerated dos
  Bortezomib: This study is designed to assess the safety, tolerance and activity of daily oral vandetanib and bortezomib on days 1, 4, 8 & 11 every 28 days in adults
  Vandetanib: This study is designed to assess the safety, tolerance and activity of daily oral vandetanib and bortezomib on days 1, 4, 8 & 11 every 28 days in adults
- Phase 2 A: Patients will be treated with vandetanib and bortezomib at the maximally tolerated dose of the Phase I study
  Bortezomib: This study is designed to assess the safety, tolerance and activity of daily oral vandetanib and bortezomib on days 1, 4, 8 & 11 every 28 days in adults
  Vandetanib: This study is designed to assess the safety, tolerance and activity of daily oral vandetanib and bortezomib on days 1, 4, 8 & 11 every 28 days in adults
- Total: Total of all reporting groups
Arm/Group | Phase 1 | Phase 2 A | Total
Number analyzed (Participants) | 21 | 1 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 1 | 17
  >=65 years | 5 | 0 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.07 (10) | 39.8 (0) | 55.34 (10.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 0 | 8
  Male | 13 | 1 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 20 | 1 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 18 | 0 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 1 | 22

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Maximum Tolerated Dose (MTD) of Daily Oral Vandetanib
Description: A maximum tolerated dose for vandetanib will be determined if dose limiting toxicity is observed in 2 or more patients at one of the dose levels being evaluated. The MTD will be the dose level immediately preceding the dose level at which DLT (e.g. defined as neutrophil count below 1000/ µL (grade 3) on 2 consecutive measurements drawn at least 72 hours OR a single neutrophil count below 500/µL occurred. Platelet count below 50,000 µL (grade 3) on 2 consecutive measurements drawn at least 72 hours apart OR a singe platelet count below 25,000/µL. A platelet transfusion administered when platelet count is below 50,000/µL is dose limiting thrombocytopenia, unless the transfusion is being administered for peri-operative coverage.
Time Frame: 80 days
Measure: Number; unit: mg
Groups:
- Phase 1: Patients will be treated with vandetanib to find the maximally tolerated dose.
  Vandetanib: This study is designed to assess the safety, tolerance and activity of daily oral vandetanib on days 1, 4, 8 & 11 every 28 days in adults
Arm/Group | Phase 1
Number analyzed (Participants) | 21
mg | 300

2. Primary Outcome: Phase I: Maximum Tolerated Dose (MTD) of Daily Oral Bortezomib
Description: A maximum tolerated dose for bortezomib will be determined if dose limiting toxicity is observed in 2 or more patients at one of the dose levels being evaluated. The MTD will be the dose level immediately preceding the dose level at which DLT (e.g. defined as neutrophil count below 1000/ µL (grade 3) on 2 consecutive measurements drawn at least 72 hours OR a single neutrophil count below 500/µL occurred. Platelet count below 50,000 µL (grade 3) on 2 consecutive measurements drawn at least 72 hours apart OR a singe platelet count below 25,000/µL. A platelet transfusion administered when platelet count is below 50,000/µL is dose limiting thrombocytopenia, unless the transfusion is being administered for peri-operative coverage.
Time Frame: 80 days
Measure: Number; unit: mg/m^2
Groups:
- Phase 1: Patients will be treated with bortezomib to find the maximally tolerated dos
  Bortezomib: This study is designed to assess the safety, tolerance and activity of daily oral bortezomib on days 1, 4, 8 & 11 every 28 days in adults
Arm/Group | Phase 1
Number analyzed (Participants) | 21
mg/m^2 | 1.3

3. Primary Outcome: Phase 2: Tumor Response in Adults With a Diagnosis of Medullary Thyroid Cancer (MTC) Treated With Daily Oral Vandetanib and Bortezomib
Description: Response is assessed by the Response Evaluation Criteria in Solid Tumors (RECIST). Complete response is disappearance of all target lesions. Partial response is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. Progressive disease is at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Stable disease is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: 4 months
Population: No participants were enrolled in the phase IIB cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 A
Number analyzed (Participants) | 1
Participants
  Complete Response | 0
  Partial Response | 0
  Stable Disease | 0
  Progressive Disease | 1

4. Primary Outcome: Phase 2: Progression Free Survival in Adults With a Diagnosis of Medullary Thyroid Cancer (MTC) Treated With Daily Oral Vandetanib and Bortezomib
Description: Progression free survival is defined as the duration of time from start of treatment to time of progression. Progression is assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) and is defined as the appearance of one or more new lesions or unequivocal progression of existing non-target lesions. Although a clear progression of "non-target" lesions only is exceptional, the opinion of the treating physician should prevail in such circumstances, and the progression status should be confirmed at a later time by the review panel (or Principal Investigator).
Time Frame: 4 months
Population: No participants were enrolled in the phase IIB cohort. One participant was in cohort 2A, thus standard deviation could not be calculated.
Measure: Median (Standard Deviation); unit: months
Arm/Group | Phase 2 A - Vandetanib and Bortezomib at the MTD
Number analyzed (Participants) | 1
months | 3.67

5. Secondary Outcome: Response Rate (Complete Response (CR) + Partial Response (PR) of Adults With a Diagnosis of MTC Treated With Either of Two Regimens: (1) Daily Oral Vandetanib and Bortezomib or (2) Daily Oral Vandetanib
Description: Comparison of response between cohorts 1, 2A and 2B was to be determined by computed tomography scan reviews using the Response Evaluation Criteria in Solid Tumors (RECIST). Complete response is disappearance of all target lesions. Partial response is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD.
Time Frame: 2-3 years
Population: A comparison between phase 1, 2A and 2B was not done because no participants were enrolled in the phase 2B cohort.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 2A: Patients will be treated with vandetanib and bortezomib at the maximally tolerated dose of the Phase I study
  Bortezomib: This study is designed to assess the safety, tolerance and activity of daily oral vandetanib and bortezomib on days 1, 4, 8 & 11 every 28 days in adults
  Vandetanib: This study is designed to assess the safety, tolerance and activity of daily oral vandetanib and bortezomib on days 1, 4, 8 & 11 every 28 days in adults
Arm/Group | Phase 1 | Phase 2A
Number analyzed (Participants) | 21 | 1
Participants
  Complete Response | 0 | 0
  Partial Response | 6 | 0

6. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression free survival is defined as the duration of time from start of treatment to time of progression. Comparison of PFS between cohorts 1, 2A and 2B was to be assessed by the Response Evaluation Criteria in Solid Tumors (RECIST). Progressive disease is at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: 2-3 years
Population: A comparison between phase 1, 2A and 2B was not done because no participants were enrolled in the phase 2B cohort.
Measure: Median (Full Range); unit: Months
Arm/Group | Phase 1 | Phase 2A
Number analyzed (Participants) | 21 | 1
Months | 30.2 [1.8 to 93.67] | 3.02

7. Secondary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE) v4.0. For the detailed list of adverse events see the adverse event module.
Time Frame: Date treatment consent signed to date off study, approximately 7 years and 9 days
Population: No participants were enrolled in the phase IIB cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 | Phase 2 A
Number analyzed (Participants) | 21 | 1
Participants | 21 | 0

8. Secondary Outcome: Number of Participants With Tumor Biomarker Calcitonin (CTN) Response
Description: Calcitonin was measured by the biomarker response criteria. Complete response (CR) is normalization (≤ upper limit of normal) of CTN level following treatment, confirmed with a repeat CTN level at least 4 weeks apart. Partial response (PR) is a ≥50% decrease in the CTN level relative to the baseline level, confirmed with a repeat CTN level at least 4 weeks apart. Progressive disease is a ≥50% increase in the CTN relative to the baseline level, confirmed with a repeat CTN level at least 4 weeks apart. Stable disease is <50% increase or decrease in CTN level relative to the baseline level.
Time Frame: 4 weeks
Population: No participants were enrolled in the phase IIB cohort. Only participants with average pre-treatment CTN levels that are >2 times the upper limit of normal are evaluable for biomarker response. There were 16 participants that met this criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 | Phase 2A
Number analyzed (Participants) | 16 | 1
Participants
  Complete response | 0 | 0
  Partial response | 5 | 0
  Stable disease | 6 | 0
  Progressive disease | 5 | 1
  No response | 0 | 0

9. Secondary Outcome: Number of Participants With Tumor Biomarker Carcinoembryonic Antigen (CEA) Response
Description: Carcinoembryonic Antigen (CEA) was measured by the biomarker response criteria. Complete response (CR) is normalization (≤ upper limit of normal) of CEA level following treatment, confirmed with a repeat CEA level at least 4 weeks apart. Partial response (PR) is a ≥50% decrease in the CEA level relative to the baseline level, confirmed with a repeat CEA level at least 4 weeks apart. Progressive disease is a ≥50% increase in the CEA relative to the baseline level, confirmed with a repeat CEA level at least 4 weeks apart. Stable disease is <50% increase or decrease in CEA level relative to the baseline level.
Time Frame: 4 weeks
Population: No participants were enrolled in the phase IIB cohort. Only participants with average pre-treatment CEA levels that are >2 times the upper limit of normal are evaluable for biomarker response. There were 14 participants that met this criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 - Vandetanib and Bortezomib | Phase 2 A
Number analyzed (Participants) | 14 | 1
Participants
  Complete response | 0 | 0
  Partial response | 2 | 0
  Stable disease | 9 | 0
  Progressive disease | 3 | 1
  No response | 0 | 0

10. Secondary Outcome: Percentage of Participants With a Change in Frequency in Tumor-Related Diarrhea Compared to Baseline
Description: Complete response is an average of 0-2 formed stools per day for a period of at least 4 weeks. partial response is a ≥50% decrease in the average stool frequency relative to baseline and a change in stool consistency from watery to loose (partially formed) for a period of at least 4 weeks. No response is criteria for CR or PR not met. Only patients with a stool frequency of ≥5/day and a stool consistency of watery will be evaluable for clinical response.
Time Frame: Baseline, and for a period of at least 4 weeks post study drug administration
Population: This outcome measure was not analyzed because no participant had a baseline diarrhea that met the criteria for analysis. They needed to have diarrhea 5 times a day for several days in a row and no one had the baseline problem.
Arm/Group | Phase 1 - Vandetanib and Bortezomib
Number analyzed (Participants) | 0

11. Secondary Outcome: Percentage of Participants With a Change in Consistency in Tumor-Related Diarrhea Compared to Baseline
Description: Baseline stool consistency (formed, loose or partially formed, watery) will be the consistency most frequently observed during a 7-day period immediately prior to starting vandetanib. Complete response (CR) is an average of 0-2 formed stools per day for a period of at least 4 weeks. Partial response (PR) is a ≥50% decrease in the average stool frequency relative to baseline and a change in stool consistency from watery to loose (partially formed) for a period of at least 4 weeks. No response is criteria for CR or PR not met. Only patients with a stool frequency of ≥5/day and a stool consistency of watery will be evaluable for clinical response.
Time Frame: Baseline, and for a period of at least 4 weeks post study drug administration
Population: This outcome measure was not analyzed because the number of patients eligible for this response is 0, in both the Phase I and Phase II cohorts. None of the participants met the criteria of >=5 watery stools per day at baseline. No participants were enrolled in the phase IIB cohort.
Arm/Group | Phase 1 - Vandetanib and Bortezomib
Number analyzed (Participants) | 0

12. Secondary Outcome: Maximum Bortezomib Plasma Concentration Normalized to Dose (Cmax/D)
Description: Geometric mean for Bortezomib pharmacokinetic (PK) parameters both before (cycle 1 day 1) and during steady-state Vandetanib (cycle 3 day 1; exposures are dose normalized). Bortezomib plasma concentrations were measured using a validated LC-MS/MS assay with a lower limit of quantification (LLOQ) of 1 ng/mL. Only measured concentrations above the LLOQ were used in the calculation of PK parameters. The maximum plasma concentration (Cmax) was recorded as observed values.
Time Frame: Cycle 1 day 1, and cycle 3 day 1 (an average of 61 days); and Pre-dose, 1, 2,4, 6, 8, 10 and 24 hours post dose
Population: "7/14 patients were analyzed on day 1; 13/14 patients analyzed on day 61. Those patients that were not analyzed had insufficient PK data to calculate this parameter."
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL/mg
Arm/Group | Phase 1 - Vandetanib and Bortezomib
Number analyzed (Participants) | 14
ng/mL/mg
  Before Vandetanib: number analyzed (Participants) | 7
  Before Vandetanib | 0.98 [0.72 to 1.24]
  After Vandetanib: number analyzed (Participants) | 13
  After Vandetanib | 1.92 [0.99 to 2.85]
Statistical Analysis 1: Comparison: Phase 1 - Vandetanib and Bortezomib; Patients given bortezomib on cycle 1, day 1 vs. cycle 3, day 1. A paired analysis among same 14 patients on Phase 1 portion. To assess whether presence of vandetanib significantly altered bortezomib Cmax (normalized to dose); Test type: Superiority or Other; p = 0.019, Mann-Whitney; (nonparametric unpaired t-test; assumed homoscedasticity)

13. Secondary Outcome: Area Under the Bortezomib Plasma Concentration Versus Time Curve From Time Zero to Infinity/Dose (AUCinf/D)
Description: The area under the concentration-time curve (AUC) extrapolated to infinity (AUCinf) was calculated using the linear up-log down trapezoidal method via extrapolation of AUC(LAST) (AUC to the last quantifiable time point) by dividing C(LAST) (the last measurable drug concentration, typically at 24 hour post-dose) by the rate constant of the terminal phase, lambda z. This constant was determined from the slope of the terminal phase of the concentration-time curve using weighted least-squares as the estimation procedure.
Time Frame: Cycle 1 day 1, and cycle 3 day 1 (an average of 61 days); and Pre-dose and 1, 2, 4, 6, 8, 10, and 24 hours post dose
Population: PK samples were only done during the phase I portion of the study. "7/14 patients were analyzed on day 1; 13/14 patients analyzed on day 61. Those patients that were not analyzed had insufficient PK data to calculate this parameter." Please see other outcome measure modules for details.
Measure: Geometric Mean (95% Confidence Interval); unit: hr*ng/mL/mg
Arm/Group | Phase 1 - Vandetanib and Bortezomib
Number analyzed (Participants) | 14
hr*ng/mL/mg
  Before Vandetanib: number analyzed (Participants) | 7
  Before Vandetanib | 1.27 [0.57 to 1.97]
  After Vandetanib: number analyzed (Participants) | 13
  After Vandetanib | 2.39 [1.67 to 3.11]
Statistical Analysis 1: Comparison: Phase 1 - Vandetanib and Bortezomib; Patients given bortezomib on cycle 1 day 1 vs. cycle 3 day 1. A paired analysis among same 14 patients on Phase 1 portion. To assess whether presence of vandetanib significantly altered bortezomib AUCinf (normalized to dose); Test type: Superiority or Other; p = 0.052, Mann-Whitney; (nonparametric unpaired t-test; assumed homoscedasticity)

14. Secondary Outcome: Terminal Half-Life (T1/2) of Bortezomib
Description: The time it takes for the measured concentration of the drug to drop by half.
Time Frame: Cycle 1 day 1, and cycle 3 day 1 (an average of 61 days); and Pre-dose and 1, 2, 4, 6, 8, 10, and 24 hours post dose
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: hour
Arm/Group | Phase 1
Number analyzed (Participants) | 14
hour
  Before Vandetanib: number analyzed (Participants) | 7
  Before Vandetanib | 9.4 [3.5 to 15.4]
  After Vandetanib: number analyzed (Participants) | 13
  After Vandetanib | 12.5 [7.3 to 17.7]
Statistical Analysis 1: Comparison: Phase 1; Patients given bortezomib on cycle 1 day 1 vs. cycle 3 day 1. A paired analysis among same 14 patients on Phase 1 portion. To assess whether presence of vandetanib significantly altered bortezomib half-life; Test type: Superiority or Other; p = 0.440, Mann-Whitney; (nonparametric unpaired t-test; assumed homoscedasticity)

15. Secondary Outcome: Total Systemic Clearance (CL) of Bortezomib
Description: Total systemic clearance = dose/area under curve extrapolated to infinity (AUCinf.). This measurement represents the rate at which plasma is systematically cleared of drug.
Time Frame: Cycle 1 day 1, and cycle 3 day 1 (an average of 61 days); and Pre-dose and 1, 2, 4, 6, 8, 10, and 24 hours post dose
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: L/hr
Arm/Group | Phase 1
Number analyzed (Participants) | 14
L/hr
  Before Vandetanib: number analyzed (Participants) | 7
  Before Vandetanib | 78.7 [37.6 to 120]
  After Vandetanib: number analyzed (Participants) | 13
  After Vandetanib | 42.9 [30.4 to 55.4]
Statistical Analysis 1: Comparison: Phase 1; Patients given bortezomib on cycle 1 day 1 vs. cycle 3 day 1. A paired analysis among same 14 patients on Phase 1 portion. To assess whether presence of vandetanib significantly altered bortezomib clearance; Test type: Superiority or Other; p = 0.016, Mann-Whitney; (nonparametric unpaired t-test; assumed homoscedasticity)

16. Secondary Outcome: Bortezomib Volume of Distribution (Vss)
Description: Vss represents the volume into which the drug distributes into once given to the patient at steady-state. This volume parameter provides a measure of where in the body the drug is going, based on fluid volume.
Time Frame: Cycle 1 day 1, and cycle 3 day 1 (an average of 61 days); and Pre-dose and 1, 2, 4, 6, 8, 10, and 24 hours post dose
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: Liter
Arm/Group | Phase 1
Number analyzed (Participants) | 14
Liter
  Before Vandetanib: number analyzed (Participants) | 7
  Before Vandetanib | 1167 [1049 to 1286]
  After Vandetanib: number analyzed (Participants) | 13
  After Vandetanib | 749 [580 to 918]
Statistical Analysis 1: Comparison: Phase 1; Patients given bortezomib on cycle 1 day 1 vs. cycle 3 day 1. A paired analysis among same 14 patients on Phase I portion. To assess whether presence of vandetanib significantly altered bortezomib volume of distribution; Test type: Superiority or Other; p = 0.010, Mann-Whitney; (nonparametric unpaired t-test; assumed homoscedasticity)

17. Secondary Outcome: Comparison of Steady State Vandetanib Exposure With Relevant Literature Values
Description: Because vandetanib PK exposure was only measured during a single 8-hr window during daily dosing, the only comparison to assess the effect of bortezomib is to compare these values to published literature."
Time Frame: Cycle 3 day 1 (an average of 60 days); and Pre-dose and 1, 2, 4, 6, 8, 10, and 24 hours post dose
Population: Vandetanib PK samples were only obtained during the phase 1 portion of the study during cycle 3, day 1, where patients received both vandetanib (at steady-state) and bortezomib. "13/14 patients analyzed on day 61 (C3D1). Those patients that were not analyzed had insufficient PK data to calculate this parameter."
Measure: Mean (Standard Deviation); unit: ng/mL/mg
Arm/Group | Phase 1 - Vandetanib and Bortezomib
Number analyzed (Participants) | 14
ng/mL/mg
  Published Literature | 4.77 (1.8)
  Study 090089 Results: number analyzed (Participants) | 13
  Study 090089 Results | 3.96 (0.89)

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 7 years and 9 days.
Description: No participants were enrolled in the phase IIB cohort.
Arm/Group | Phase 1 | Phase 2 A
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/1
Serious Adverse Events (participants affected / at risk) | 4/21 | 1/1
Other Adverse Events (participants affected / at risk) | 21/21 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 (N=21) | Phase 2 A (N=1)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (2) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 (N=21) | Phase 2 A (N=1)
Abdominal pain (Gastrointestinal disorders) | 7 (16) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 3 (6) | 0 (0)
Alanine aminotransferase increased (Investigations) | 20 (72) | 1 (1)
Alkaline phosphatase increased (Investigations) | 4 (10) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 9 (31) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 5 (5) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 19 (61) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 3 (3) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Bronchial infection (Infections and infestations) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
CPK increased (Investigations) | 5 (10) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (4) | 0 (0)
Chills (General disorders) | 5 (7) | 0 (0)
Constipation (Gastrointestinal disorders) | 8 (12) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 1 (1)
Creatinine increased (Investigations) | 7 (22) | 1 (2)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 3 (4) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 16 (78) | 0 (0)
Dizziness (Nervous system disorders) | 4 (7) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 7 (9) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphasia (Nervous system disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Edema limbs (General disorders) | 2 (6) | 0 (0)
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 19 (93) | 1 (2)
Eye infection (Infections and infestations) | 2 (2) | 0 (0)
Eyelid function disorder (Eye disorders) | 3 (3) | 0 (0)
Fatigue (General disorders) | 13 (37) | 0 (0)
Fever (General disorders) | 5 (7) | 0 (0)
Flushing (Vascular disorders) | 1 (3) | 0 (0)
GGT increased (Investigations) | 4 (4) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 6 (7) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hemoglobinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 0 (0)
Hot flashes (Vascular disorders) | 2 (3) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 4 (5) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (6) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5 (12) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 8 (11) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 11 (28) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 7 (8) | 0 (0)
Hypertension (Vascular disorders) | 15 (24) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 2 (2) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 19 (98) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 11 (22) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 3 (17) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 6 (19) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 10 (22) | 1 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 5 (8) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 5 (6) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 6 (7) | 0 (0)
Investigations - Other, specify (Investigations) | 5 (9) | 0 (0)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 2 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 20 (121) | 1 (2)
Mucositis oral (Gastrointestinal disorders) | 2 (2) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (7) | 0 (0)
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nail loss (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 13 (21) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (2)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 2 (6) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (5) | 0 (0)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 4 (7) | 0 (0)
Pain in extremity (General disorders) | 2 (2) | 0 (0)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 4 (6) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Peripheral nerve infection (Infections and infestations) | 2 (2) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 11 (17) | 0 (0)
Photosensitivity (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0)
Platelet count decreased (Investigations) | 17 (93) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 11 (34) | 1 (2)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 10 (20) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9 (15) | 0 (0)
Renal calculi (Renal and urinary disorders) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 3 (4) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 2 (3) | 1 (1)
Sinusitis (Infections and infestations) | 2 (3) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Skin infection (Infections and infestations) | 2 (2) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (2) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (4) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Weight loss (Investigations) | 4 (6) | 1 (1)
White blood cell decreased (Investigations) | 12 (46) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2015-08-18): https://cdn.clinicaltrials.gov/large-docs/47/NCT00923247/Prot_000.pdf